CLINICAL TRIAL: NCT04506476
Title: Randomisierte Studie Zum Nutzen Des Fitnesstracker Basierten Aktivitätstrainings während Einer Adjuvanten Bestrahlung Des Mammakarzinoms (OnkoFit I)
Brief Title: Trial Evaluating the Benefit of a Fitness Tracker Based Workout During Adjuvant Radiotherapy of Breast Cancer
Acronym: OnkoFit I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Cihan Gani, Senior Physician, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OnkoFit I
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
Keywords: Fatigue; activity tracker; Radiotherapy; Exercise
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Activity tracker with weekly goals (Experimental): Patients receive a fitness tracker, a booklet "Physical training, exercise and cancer" and an in-person briefing on physical activity during cancer therapy. We suggest a daily step-count which should improve the patients physical activity during radiotherapy of breast cancer. Patients receive weekly feedback and a new goal with the aim to reach a total of 6000 daily steps, which should be then maintained during radiotherapy.
  Interventions: Device: Fitness tracker based activity training for Arm A and B. Booklet "physical training, exercise and cancer" and an introduction about physical activity during cancer therapy for Arm A, B, C
- Activity tracker without Weekly goals (Experimental): Patients receive a fitness tracker, a booklet "Physical training, exercise and cancer" and an in-person briefing on physical activity during cancer therapy.
  The patients self-document their daily step count during radiotherapy, there will be no recommendation for the daily count of steps.
  Interventions: Device: Fitness tracker based activity training for Arm A and B. Booklet "physical training, exercise and cancer" and an introduction about physical activity during cancer therapy for Arm A, B, C
- Control arm with no activity tracker (No Intervention): Patients receive a booklet "Physical training, exercise and cancer" and an in-person briefing on physical activity during cancer therapy. A fitness tracker will not be provided.

INTERVENTIONS:
Device: Fitness tracker based activity training for Arm A and B. Booklet "physical training, exercise and cancer" and an introduction about physical activity during cancer therapy for Arm A, B, C — Patients receive a fitness tracker, a booklet "Physical training, exercise and cancer" and an in-person briefing about physical activity during cancer therapy. With offered guidelines for the daily step counts patients should improve their physical activity during radiotherapy of breast cancer. A weekly feedback and a new goal for the next week will be provided until the individual patient reaches a daily activity of 6000 steps. The setting will be to maintain to this daily activity of 6000 steps during radiotherapy.
  Arms: Activity tracker with weekly goals; Activity tracker without Weekly goals

SUMMARY:
This randomized three-arm trial will test the benefit in terms of cancer related fatigue of an activity tracker based exercise training during adjuvant radiotherapy in breast cancer patients.

DETAILED DESCRIPTION:
This monocentric, three-arm, randomized, controlled clinical trial evaluates the effect of an activity tracker based exercise program in breast cancer patients on the fatigue syndrome during adjuvant radiotherapy. Quality of Life and the intensity of fatigue will be documented with the fatigue subscale of the FACIT Questionnaire three months after adjuvant radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Capacity for consent
* Minimum age 18
* Presence of breast cancer
* ECOG 0-2
* Indication for adjuvant radiotherapy of breast cancer after breast-conserving surgery or Ablatio mammae

Exclusion Criteria:

* Participation in any other interventional study
* Pregnancy
* Contraindication against physical activity/sport and others
* Severe cardiovascular pre-existing conditions (after myocardial infarction, apoplexy in the last 6 months, congestive heart failure NYHA > I°)
* preexisting diseases with are relevantly accompanied by a limited mobility in patients (e.g. paraparesis of the lower limbs)
* ECOG Status 3-4
* prior use of activity trackers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the impact of an activity tracker based fitness programme on the fatigue syndrome | 3 Months after completion of adjuvant radiotherapy of breast cancer
  This endpoint will be evaluated by the FACIT-F (Functional Assessment of Chronic Illness Therapy-Fatigue) subscale of the FACIT questionnaire (Physical well-being values 0-28, 28 worse outcome; social/family well-being values 0-28, 28 better outcome; emotional well-being values 0-24, 24 worse outcome; functional well being values 0-28, 28 better outcome; additional factors values 0-64, 64 worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Gani, MD, PD, Principal Investigator — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Department of Radiation Oncology, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Hauth F, Gehler B, Niess AM, Fischer K, Toepell A, Heinrich V, Roesel I, Peter A, Renovanz M, Hartkopf A, Stengel A, Zips D, Gani C. An Activity Tracker-Guided Physical Activity Program for Patients Undergoing Radiotherapy: Protocol for a Prospective Phase III Trial (OnkoFit I and II Trials). JMIR Res Protoc. 2021 Sep 22;10(9):e28524. doi: 10.2196/28524. PMID 34550079